CLINICAL TRIAL: NCT03784313
Title: Secondary Intention Wound Healing Versus Axillary Perforator Flaps for Axillary Reconstruction, After Surgical Wide Excision for Hidradenitis Suppurativa : a Randomized Multicentered Controlled Trial
Brief Title: Perforator Flaps for Axillary Hidradenitis Suppurativa
Acronym: HS-PAX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P170931J; 2018-A01244-51 (Other: ANSM)
Record Dates: First submitted 2018-11-13; First posted 2018-12-21 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Axillary Hidradenitis Suppurativa
Keywords: Axillary Hidradenitis Suppurativa; Perforator flaps; Secondary intention wound healing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perforators flaps (PF group) (Experimental)
  Interventions: Procedure: skin repair by axillary perforator flaps
- Secondary intention wound healing (Sham Comparator)
  Interventions: Procedure: skin repair by secondary wound healing

INTERVENTIONS:
Procedure: skin repair by axillary perforator flaps — Perforators flaps (PF) of the axillary region for the coverage the axillary defect left after radical excision for axillary Hidradenitis Suppurativa.
  Perforated flap surgery does not involve any procedure or manipulation that may alter the biological characteristics and/or structural properties of the tissue (use autologue pur). A usual dressing is performed daily until complete healing.
  Arms: Perforators flaps (PF group)
Procedure: skin repair by secondary wound healing — Secondary intention wound healing (SIWH) for the coverage the axillary defect left after radical excision for axillary Hidradenitis Suppurativa
  Arms: Secondary intention wound healing

SUMMARY:
Hidradenitis Suppurativa (HS) is a recurrent inflammatory disease (< 2 episode /6 months) with 1%-4% prevalence in Europe. Suppurating lesions are painful and involve one or more regions (axilla, genitofemoral, perineum, gluteal areas and inframammary, creases).

For recalcitrant stage II and III, wide surgical skin excision is the only recommended and validated treatment in case inefficacity of medical conventional systemic therapies or limited-local surgery.

Perforator Flaps (PF) surgery, are a new and innovative surgical technique, that, unlike secondary wound healing, allows a single stage reconstruction at the same time as skin excision without its disadvantages.: prolonged healing time, with multiple painful dressings (costs) retractile scar with reduction of the range of motion, dyschromia, unstable and fragile scar.

The hypothesis of study is a 30% reduction of time to healing by using perforators flaps technique (PF) versus wound healing (SIWH), for axillary reconstruction after surgical wide excision in axillary hidradenitis suppurativa stage II or III in adults with inadequate response to conventional systemic therapy.

DETAILED DESCRIPTION:
This study is designed as an open randomized clinical trial comparing the efficacy of perforators flaps technique (PF) to decrease the healing time, versus secondary intention wound healing (SIWH) after skin excision for axillary Hidradenitis suppurativa.

This study involves 8 centers (2 closed) plastic surgery

Patients will be randomized by the investigator after inclusion using a Case Report Form (e-CRF) CleanWeb, Telemedecin Technologies, S.A.S). Randomization will be stratified on center and on laterality (unilateral/bilateral); in case of bilateral axillary HS, side will be randomly assigned at the same time than surgery group.

Centralized blocked randomization according to a 1:1 ratio will be prepared by the Clinical Research Unit (URC-EST).

Primary endpoint

Healing time defined as :

1. In SIWH group: time between the excisional surgery and total re-epithelialization (100%), treatment of potential wound healing delay related to complications included.
2. in PF group : time between the excisional surgery and the day of last stiches removal(closed incision), treatment of potential delay related to complications included .If partial necrosis< 50 %, occurs and is treated by SIWH , the secondary end point will be the total re-epithelialization.

If healing is not attended at the end of follow up, healing duration will be set at 6 months in both group

Secondary endpoints

To compare between groups:

* Recurrence rate during a follow-up of 12 months: new signs of disease in the axilla despite surgical treatment and Hurley staging of the involved axilla .
* Disabilities of the Arm, Shoulder and Hand score (DASH) and of the measurement of the amplitude of arm abduction using a goniometer : differences between inclusion and M3, M6, M12.
* Length of stay at the hospital at the discharge
* Time from surgery to return to daily activity
* Quality of life between inclusion and at M3, M6, M12; with MOS-SF36 / Dermatology Life Quality Index (DLQI)/ EQ 5D
* Aesthetic outcomes: VAS (1: worst aesthetic result-10 : best aesthetic result) obtained after submission of the pre/post-operative pictures of the axillary region to a medical/paramedical panel at M12 and patient satisfaction for the aesthetic outcomes at M12 with the same scale, Pre/post-operative pictures of the axillary region will be submitted to a medical/paramedical panel and measured with the same Visual Analogic scale (VAS) aesthetic outcomes 3 Pictures
* 1 face Arm elevated with the 2 axillae in the frame, 1 of the axillae face, 1 of the axillae profil
* The day of the surgery or one day before surgery: a picture to determine the size of the lesion (arm 90°) and with the size of the defect (Ruler or dimension written on the skin) after skin excision.

VAS patient satisfaction for the aesthetic outcomes

* Complication rates during a follow up of 3 months: hematoma, infection, cutaneous necrosis
* Pain (Visual Analogic Scale): before patient discharge, every 15 days until wound healing and at M3 and M6.
* Production costs of the new technique perforator flap from the hospital perspective
* Total average cost and incremental cost-utility ratio

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 70 years
* Reproductive age patient with an effective contraception
* Patient with a previously diagnosed of axillary HS (defined by European S1 guidelines) Hurley Grade II or grade III and send by dermatologist for wide excision surgery, because of inefficacy, or insufficient response or failure (recurrence or resistance) of previous medical conventional systemic treatments or limited surgery
* Minimum delay of 1 month after an inflammatory phase of axillary HS treated medically
* Patient candidate for excision surface of the axillary region representing a minimum excision area of 6 (major axis) / 6 (minor axis) or 28.5 cm2 (ellipse surface recall = half of major axis X half of minor axis X π, in this case = 3 X 3 X π)
* Patient with health insurance (AME excepted)
* Signed written informed consent

Exclusion Criteria:

* Contra indication to general anesthesia, allergy to methylene blue (mandated for the excisional surgery)
* Pregnancy woman (confirmed by a urine test beta-HCG) or breastfeeding woman
* Patient already included in the study
* Participation in any other interventional study or in the exclusion period any other interventional study
* Contra indication to perforator flaps/wide excision : to general anesthesia (ASA < IV Score Health Status), severe platelet disorders or patient at high risk of bleeding
* Acute superinfection grade ≥ 4 according to CTCAE in progress or diagnosed for less than 1 month
* Patient under legal protection measure and or deprived of freedom
* Patient unable to consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2024-03-26 (Estimated); Study Completion 2024-09-24 (Estimated)

PRIMARY OUTCOMES:
To compare the efficacy at 6 months on the healing time of perforators flaps and secondary intention wound healing after wide surgical excision, for axillary HS stage II or III insufficiently responsive to conventional systemic treatment. | 6 months
  Primary assessment criterion is the mean Healing time during a 6 months follow up defined as :
  * In SIWH group: time between the excisional surgery and total re-epithelialization (100%), treatment of potential delay related to complications included.
  * in PF group : time between the excisional surgery and the day of last stiches removal(closed incision of the recipient site and donor site), treatment of potential delay related to complications included.

SECONDARY OUTCOMES:
Recurrence rate during the 12-months follow-up defined as: new signs of disease in the axilla despite surgical treatment and Hurley staging of the involved axilla | 12 months
  The recurrence severity is described by the Hurley staging of the involved axilla. Hurley staging of the involved axilla will be described and compared between groups by a Fischer's exact test.
Shoulder mobility on the operated side, evaluated by the DASH score | Day10, Month 3, Month 6 and Month12
  The DASH score (Disabilities of the Arm, Shoulder and Hand)
Shoulder mobility on the operated side, by the measurement of the amplitude of arm abduction | Day10, Month 3, Month 6 and Month12
  The amplitude of arm abduction using a goniometer
Length of stay at the hospital from surgery to the discharge | Day 7
  Length of stay at the hospital will be compared between groups using Student t tests or Wilcoxon rank-sum tests, as needed
Time from surgery to return to daily activity | Month 1, Month 3, Month 6
  Time from surgery to return to work, to school-university, daily activity (if unemployed) will be compared between groups using Student t tests or Wilcoxon rank-sum tests, as needed
Evolutions during the 12-months follow in quality of life by using MOS-SF36 | Up to Month 12.
  MOS-SF36 questionnaire will be analyzed according to the scoring manual.
Evolutions during the 12-months follow in quality of life by using DLQI | Up to Month 12.
  DLQI questionnaire will be analyzed according to the scoring manual.
Evolutions during the 12-months follow in quality of life by using EQ 5D | Up to Month 12.
  EQ5D questionnaire will be analyzed according to the scoring manual.
Aesthetic outcomes of the axillae at 12 months | Month 12
  Aesthetic outcomes at 12 months according to patients and to the medical panel (VAS 0: worst aesthetic result - 10 : best aesthetic result) will be assessed using Student t tests or Wilcoxon rank-sum tests, as needed.
Complication rates at 3 months | 3 months
  described by complication (hematoma, hemorrhage, infection, wound dehiscence, skin necrosis, scar retraction) and as a total complication rate and compared between groups using a Pearson Chi square test or a Fisher's exact test, when appropriate.
Evolution of the Analogic Visual Scale for Pain | Day10 / Day0 to Day7, Day15 Month 1/Month 3 /Month 6
  Pain evolution will be described graphically and may be compared between groups using a linear mixed model, if possible. In case of non-normality distribution of the interest variable, a transformation could be realized.
  VAS ( 0 : none 10: extreme amount of pain)
Evolution of patient satisfaction by VAS | Month 1/ Month 3/ Month 6/ Month 12
  Satisfaction evolution will be described graphically and may be compared between groups using a linear mixed model, if possible. In case of non-normality distribution of the interest variable, a transformation could be realized.
  VAS ( 0 : Totally dissatisfied 10 : Fully satisfied)
Production costs of the new technique perforator flap from the hospital perspective | 12 months
Total average cost and incremental cost-utility ratio | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael ATLAN, PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service PREMIER ( Plastique, Reconstruction, Esthétique, Microchirugie et Régénération tissulaire)CHU TENON- APHP, Paris, France

IPD SHARING:
Plan to Share IPD: No